CLINICAL TRIAL: NCT06915649
Title: Exploration and Evaluation of Amygdalo-Hippocampectomy According to Prof. Coubes' Technique: An Anatomical, Clinical, and Educational Approach
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-08-115
Record Dates: First submitted 2025-01-16; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hippocampal Sclerosis; Dysembryoplastic Neuroepithelial Tumor; Cortical Dysplasia; Ganglioglioma; Cavernoma; Epidermal Cyst; Hamartoma; Pilocytic Astrocytoma; DGONC
Keywords: hippocampal sclerosis; hippocampectomy; amygdala-hippocampectomy; epilepsy surgery
MeSH Terms: conditions — Hippocampal Sclerosis; Malformations of Cortical Development; Ganglioglioma; Hemangioma, Capillary; Epidermal Cyst; Hamartoma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients operated: We studied all the patients who underwent an Amygdalo-Hippocampectomy in the University Hospital of Montpellier, France from 1995 until 2022
  Interventions: Procedure: Amygdalo-Hippocampectomy

INTERVENTIONS:
Procedure: Amygdalo-Hippocampectomy — This technique is characterized by specific hallmarks that distinguish it from other approaches, including the Yasargil technique and newer minimally invasive methods. It integrates precise anatomical targeting with optimized surgical pathways to enhance outcomes in patients with those pathologies. The approach of the choroidal fissure will be explained in the article.
  By addressing limitations observed in traditional techniques, it aims to minimize neurological deficits while achieving better seizure control.

SUMMARY:
The goal of this retrospective study is to evaluate the long-term clinical outcomes and complications associated with amygdalo-hippocampectomy using the surgical technique developed by Pr. Coubes (Montpellier, FRANCE). The main questions it aims to answer are:

* What are the complications and evolution of clinical outcomes in patients treated with this technique for hippocampal sclerosis or other intern temporal diseases ?
* What variables are associated with better seizure control following surgery?

Participants include 234 patients treated over the last 30 years at the CHU de Montpellier, FRANCE. The study will analyze clinical data, including seizure outcomes based on ILAE criteria, post-operative complications, and factors influencing recovery and reintegration into daily life.

DETAILED DESCRIPTION:
Title Exploration and Evaluation of Amygdalo-Hippocampectomy Using Pr. Coubes' Technique: An Anatomical, Clinical, and Pedagogical Approach

Introduction The hippocampus, a vital component of the limbic system, plays a key role in memory and emotions. Unfortunately, it is also prone to various pathologies, such as hippocampal sclerosis, a condition characterized by progressive neuronal degeneration and subsequent fibrosis of the medial temporal lobe. Other diseases may occur such as tumours, Dysembryoplastic Neuroepithelial Tumour (DNET) or gliomas.

This condition often leads to severe symptoms, including pharmacoresistant epilepsy and memory disturbances that significantly impair the quality of life.

For patients with pharmacoresistant epilepsy associated with hippocampal sclerosis, surgery has emerged as a first-line therapeutic option. Among the surgical techniques, hippocampectomy and amygdalo-hippocampectomy aim to remove the affected portion of the hippocampus, reducing seizure propagation and improving patient outcomes. However, these procedures are marked by significant variability in their operative techniques, extents of resection, and patient selection criteria.

While the amygdalo-hippocampectomy technique described by Pr. Yasargil in 1985 remains a cornerstone in surgical approaches, other methods such as the trans-sylvian approach (Adada et al., 2008), the trans-gyral approach (Mathon & Clemenceau, 2016), and emerging endoscopic techniques (H. Westley Phillips, 2023) highlight the diversity and evolution of surgical options.

This study seeks to explore in detail the surgical technique developed by Pr. Coubes, analyzing its anatomical, surgical, and clinical aspects. Additionally, it aims to compare this method with other surgical approaches to understand its benefits and limitations better in managing hippocampal sclerosis.

Objectives Primary Objective

- To describe the complications and the evolution of clinical outcomes in patients treated with Pr. Coubes' amygdalo-hippocampectomy technique.

Secondary Objective - To identify variables associated with favorable seizure control and overall clinical outcomes.

Study Design Type of Study

- Retrospective, single-center study conducted at the CHU de Montpellier.

Population

* 234 patients treated with this technique between 1980 and 2023, representing over three decades of clinical practice.
* Inclusion of both adult and pediatric patients.

Data Collection

* Retrospective extraction of clinical, imaging, and surgical data from patient records via the informatic patients' system.
* Data categories include demographic details, pre- and post-operative imaging (MRI), seizure frequency and type (ILAE criteria), complications, return-to-work rates, and social reintegration metrics.

Methodology Statistical Analysis

* Kaplan-Meier survival curves : Used to evaluate the time to the occurrence of complications or changes in clinical outcomes.
* Cox proportional hazards models : Conducted in both univariate and multivariate settings to identify predictors of post-operative outcomes and complications.

Outcome Measures

* Primary outcome : Seizure control evaluated using ILAE classification.
* Secondary outcomes : Post-operative complications, return-to-work rates, and functional reintegration.

Ethical Considerations

* Data Privacy : All patient data will be pseudonymized according to the French Ethic guidelines, with storage on secure CHU servers for a maximum of two years post-publication.
* Patient Notification : Informational letters will be sent to patients, detailing the study's objectives and their rights to non-opposition.

Expected Contributions

1. Clinical Insights : Comprehensive analysis of over 30 years of surgical practice, offering robust data on the efficacy and safety of Pr. Coubes' technique.
2. Comparative Perspective : Enhanced understanding of how this technique compares to other established and emerging surgical approaches.
3. Pedagogical Value : Detailed anatomical and surgical documentation to guide future training and clinical practice in neurosurgery.

Conclusion This study represents a unique opportunity to document and analyze a long-practiced yet unpublished surgical technique. By consolidating decades of clinical experience and integrating advanced analytical methods, it aims to provide valuable insights for improving the management of hippocampal sclerosis, ultimately advancing patient care and surgical education.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone an Amygdalo-Hippocampectomy according to the surgical procedure that we describe

Exclusion Criteria:

* Patients who did not have this exact procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients that have been followed in the University Hospital of Montpellier, France in the Epileptic Ward.
Sampling Method: Non-Probability Sample
Enrollment: 3504 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Post-Surgical Classification assessing epilepsy's control | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to twenty years. The study starts in 2024 and ends in 2025, which lasts one year.
  The ILAE post-surgical classification system is used to categorize seizure outcomes after epilepsy surgery. It provides a standardized way to evaluate how effectively surgery controls seizures, enabling consistency in reporting and comparison of surgical outcomes across studies and clinical settings.
  In those cases of drug-resistance epilepsy, we will assess the epilepsy's control after the surgery.
  1. Completely seizure free; no auras
  2. Only auras; no other seizures
  3. One to three seizure days per year
  4. Four to 12 seizure days per year
  5. Daily seizures
  6. More than 100% increase of baseline ; auras

SECONDARY OUTCOMES:
Post-operative complications : Infections | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to twenty years. The study starts in 2024 and ends in 2025, which lasts one year
  Each post-operative complications have been studied during the medical follow-up. It included the immediate post-operative complications such as presence of an infection.
Post-operative complications : Hematomas | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to twenty years. The study starts in 2024 and ends in 2025, which lasts one year.
  Each post-operative complications have been studied during the medical follow-up. It included the immediate post-operative complications such as presence of hematoma.
Post-operative way of life | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to twenty years. The study starts in 2024 and ends in 2025, which lasts one year.
  As part of this research on the surgery, the investigators are studying the post-surgical way of life of patients who have undergone this procedure. This includes evaluating various aspects of their daily functioning, such as autonomy, cognitive and psychiatric outcomes, social integration, and overall quality of life. By analyzing these factors, the investigators aim to better understand the long-term impact of hippocampectomy and identify potential areas for improving patient care and rehabilitation strategies.
Risk factors or predisposing factors of success or failure after Amygdalo-Hippocampectomy | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to twenty years
  Among the patients who underwent favourable and unfavourable evolutions, we will assess the risk factors and the predisposing factors such as febrile seizure, medical history, etiologic lesions.
Anti-Seizures Medications (ASM) evolution after the surgery | Medication prescribed before the surgery and medication prescribed at the last medical follow-up, assessed up to twenty years
  The investigators have also compared the potential evolution of the medications after the surgery given the drug-resistance profil of these patients.
  The number of tablets have been reported before the surgery and at the last medical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan POULEN, MD, PhD, Study Director — CHU de MONTPELLIER, FRANCE
Locations (1):
- CHU de Montpellier, Montpellier, Hérault, France